Validation of Expert

Dear Experts:

Thank you kindly for giving your time in your busy schedule to support my research, my

name is Ai Mengqi, I am a PhD student at Universiti Putra Malaysia, major in Physical

Education, my research is under the supervision of Prof. Soh Kim Geok, my dissertation is

titled "Effect of plyometric training on lower limbs explosive strength and skill performance

among university student Latin dancer in China". I'm working on my protocol right now,

with your comments and feedback being very important to me. You are a scholar with rich

theoretical knowledge and practical experience, I cordially invite you to make suggestions for

my protocol, and I will refine and improve my protocol according to your suggestions, which

can make my experiments more reliable and can help me to continue the next step of my

research. What you fill in will be used as research material only and I will keep it absolutely

confidential and will not divulge it to anyone else. So please feel free to fill in the details.

Thank you very much for your help and cooperation!

Universiti Putra Malaysia

Supervisor committee: Prof. Dr. Soh Kim Geok

Dr. Borhannudin Bin Abdullah

| Expert Name: | Discipline: | _ |
|--------------|-------------|---|
| Degree: | Work Unit: | |

#### 1 Study Overview

### 1.1 Brief Summary

Physical fitness training improves the physical fitness level of dancers and increases their explosive power(Angioi et al., 2012; de la Cruz-Torres et al., 2019; Dowse et al., 2020; Hutt & Redding, 2014; Karim et al., 2019; Kim et al., 2017; Ko et al., 2020; Kolokythas et al., 2022; Koutedakis et al., 2007; Koutedakis & Sharp, 2004; Liu & Wang, 2024; Marshall & Wyon, 2012). In the past, traditional training methods were generally used to improve the strength of dancers, but there are drawbacks to this training method, which cannot fully develop physical fitness and may lead to athletic injuries or limitations in improving skills(Moro et al., 2020). Plyometric training is a high-intensity training method that has been shown to have significant benefits in terms of increasing explosive power (Huang et al., 2023; Ramírez-Campillo et al., 2014; Ramírez-Campillo et al., 2013). However, there is little research on the effects of plyometric training on explosive power and skill in dance programs. Exercise improves physical fitness, plyometric training improves explosive power, and plyometric training should also improve explosive power and specialized performance in Latin dancers. Therefore, the research on improving the explosive power of Latin dancers' lower limbs through plyometric training is of great theoretical and practical significance, which can find suitable means of explosive power training for Latin dance programs, provide reference for coaches in training, and increase the theoretical research on the effect of plyometric training on explosive power.

### 1.2 Detailed Description

The Intervention Protocol of this research used part of the research protocol of Chinese scholar Du Min (Du, 2020). This research utilized augmentative training as an intervention, with the dependent variables being the subject's lower limb explosive power and Latin dance skill performance. Through extensive literature review, countermovement jumps, standing long jump, and 20m-sprint were identified as measures of lower limb explosive power(Chen et al., 2023). The experimental and control groups will be tested on the same Cha Cha Dance Gold Medal solo routine and recorded with a video camera. Score athletic performance according to 'the Latin Dance Technical Quality Elements of the World DanceSport Federation (WDSF) 2.1 Evaluation System'. Lower limb explosive power is closely related to the skill performance of cha-cha dance, and the review of the relevant literature was

determined to be posture, balance, footwork, preparation-movement-reduction, spinning and rotation, dynamic performance, and line extension as the test indicators of elementary skill (pei, 2023). In order to make the experiment more rigorous and scientific, to reduce the interference of uncontrollable factors, this research is Cluster Randomized Controlled Trial (CRCT) design, the students come from different areas. This experiment lasted for 8 weeks, 1.5 hours each time (Du, 2020), including one hour of physical fitness training and half an hour of specialized technical training. The sample was a population of university students who had been studying Latin dance for one year as well as more than one year, from Guangxi Normal University (Guilin) and Guilin University of Electronic Technology (Beihai), a total of 48 people. Dancers were randomly assigned to two different training locations and divided into experimental and control groups. Both groups will be trained in the Cha Cha Dance Single Gold Medal Moves. The experimental group will undergo plyometric training and the control group will undergo general training. This study measured the dependent variable three times throughout the intervention: baseline before the experimental intervention, post-test 1 after 4 weeks, and post-test 2 after 8 weeks. Finally, statistical analysis was conducted on the three test results.

### 2 Protocol Design

The experiment will last a total of 8 weeks in order to familiarize the experimenter with the plyometric training protocol and to make the whole process more fluid. It is necessary to ensure correct technique during the jumping exercises to minimize the occurrence of injuries. This research will monitor heart rate to ensure that the training load is the same for the experimental group (plyometric training) and the control group (general training). Both groups will have the same heart rate for each session of training load from the preparation phase - training phase - stretching and relaxation phase during the intervention. The experimental and control groups will undergo 3 interventions a week, with one session lasting 90 minutes. The experimental group will perform 15 minutes of dynamic stretching, 30 minutes of Latin dance-specific technique training, 30 minutes of plyometric training, and 15 minutes of relaxation stretching. The control group will perform 15 minutes of general training, and 15 minutes of relaxation stretching.

**Table 1 Training Intervention Information** 

| Week | Frequency | Types | Duration (min) | Warm -up<br>/min | Physical training /min | Specialized Training | Cool-down<br>/min | Intensity | Suggestions |
|---|---|---|---|---|---|---|---|---|---|
| 1-3 | 3times/week | Plyometric<br>Training | 90min | 15min | 30min | 30min | 15 | (40%-50%)<br>HRmax | |
| | | General<br>Training | | | | | | (60%-70%)<br>HRmax | |
| 4-5 | 3times/week | Plyometric<br>Training | 90min | 15min | 30min | 30min | 15 | (60%-70%)<br>HRmax | |
| 4-3 | Junes/ Week | Standard<br>Training | John | 1311111 | Johnn | John | | (60%-70%)<br>HRmax | |
| 6-8 | 3times/week | Plyometric<br>Training | 90min | 15min | 30min | 30min | 15 | (80%-90%)<br>HRmax | |
| | Junies/ Week | Standard<br>Training | ) J | 1011111 | 5,1111 | 5 5 | | (70%-85%)<br>HRmax | |

**Table 2 Plyometric Training Protocol for Experimental Group** 

| Week | Movements | Sets/reps | Rest (sets/reps) | Intensity | Warm up | Cool down |
|---|---|---|---|---|---|---|
| | Standing Vertical Jump Consecutive leapfrog | 10sets / 3reps 8sets / | | | | |
| | Squat jump | 2reps<br>6sets /<br>3reps | | (40%-50%) | Move the wrist, | Muscle stretching— arm cross stretch, |
| 1-3 | Rocket jump | 6sets /<br>3reps | 60-120s | HRmax | shoulder,<br>hip, knee, | low lunge stretch, half split, ankle to knee |
| | High knee | 10sets /<br>3reps | | | and ankle. | ankle to knee |
| | Jumping jacks<br>followed by<br>lateral quick run | 10sets /<br>2reps | | | | |
| | Jump on the jump box Frontal consecutive | 10sets /<br>3reps<br>8sets / | | | | |
| | jumping obstacle | 3reps | | | | Muscle stretching—<br>arm cross stretch,<br>low lunge stretch, |
| 4.5 | Rocket jump | 10sets /<br>3reps | 60 120 | (60%-70%) | Move the wrist, shoulder, hip, knee, and ankle. | |
| 4-5 | Star jump | 6sets /<br>3reps | 60-120s | HRmax | | half split,<br>ankle to knee |
| | Squat jump | 10sets /<br>3reps | | | and anxic. | |
| | Consecutive | 6sets / | | | | |
| | leapfrog Tuck jump | 3reps<br>10sets /<br>3reps | | | | |
| | Weighted leapfrog followed by vertical jump | 10sets /<br>3reps | | | Move the | |
| | Jump on the jump box | 10sets /<br>3reps | 60.100 | (80%-90%) | wrist, | Muscle stretching—<br>arm cross stretch, |
| 6-8 | Depth jump followed by jump on the jump box | 8sets /<br>3reps | 60-120s | HRmax | shoulder,<br>hip, knee,<br>and ankle. | low lunge stretch,<br>half split,<br>ankle to knee |
| | Depth jump over | 10sets / | | | | |
| | obstacle Side lunge | 3reps<br>10sets /<br>3reps | | | | |

**Table 3 General Training Protocol for Control Group** 

| Week | Movements | Sets/reps | Rest (sets/reps) | Intensity | Warm up | Cool down |
|---|---|---|---|---|---|---|
| | Jumping Jacks | 15sets /<br>3reps | | | | Muscle<br>stretching—<br>arm cross stretch, |
| | Split-legged<br>left-right jump | 10sets /<br>3reps | | | Move the | |
| 1.2 | 50%1RM squat | 10sets /<br>3reps | 60.120- | (60%-70%) | wrist,<br>shoulder, | |
| 1-3 | Single-leg squat | 10sets /<br>3reps | 60-120s | HRmax | hip, knee,<br>and ankle. | low lunge stretch, half split, |
| | Supine leg raise | 10sets /<br>3reps | | | | ankle to knee |
| | Horizontal skip | 10sets /<br>3reps | | | | |
| | 20%1RM Calf<br>raises | 10sets /<br>3reps | | | | |
| | 60%1RM Squat | 10sets /<br>3reps | 60.120 | | <b>N</b> 1 | Muscle |
| | 50%1RM<br>Deadlift | 10sets /<br>3reps | | (60%-70%) | Move the wrist, | stretching—<br>arm cross stretch, |
| 4-5 | Split-legged left-right jump | 10sets /<br>3reps | 60-120s | HRmax | shoulder,<br>hip, knee, | low lunge stretch, half split, |
| | Horizontal skip | 10sets /<br>3reps | | | and ankle. | ankle to knee |
| | Lunge squat | 10sets /<br>3reps | | | | |
| | 30%1RM Calf<br>raises | 10sets /<br>3reps | | | | |
| | 60%1RM squat | 10sets /<br>3reps | | | <b>N</b> 1 | Muscle |
| 6.0 | 50%1RM<br>Deadlift | 10sets /<br>3reps | 60.120 | (70%-85%) | Move the wrist, | stretching—<br>arm cross stretch, |
| 6-8 | Lunge squat | 10sets /<br>3reps | 60-120s | HRmax | shoulder,<br>hip, knee, | low lunge stretch, half split, |
| | Standing leg lift | 15sets /<br>3reps | | | and ankle. | ankle to knee |
| | Prone sprint | 30sets /<br>3reps | | | | |

# 3 Questionnaire information

The questionnaire adopts a 4-point ordinal scale to evaluate intervention, with 1-4 representing increasing support (1=not relevant, 2=somewhat relevant, 3=quite relevant, 4=highly relevant). Please score the plyometric training intervention. If there are other content, you can add them and indicate the name. After reading the questionnaire, please rate the following aspects and tick " $\sqrt{}$ "on the corresponding rating scale.

**Table 4 Expert Evaluation Form** 

| Time | | Relevance | | | | Cl | arity | Improvement suggestions | |
|---|---|---|---|---|---|---|---|---|---|
| Туре | 4 | 3 | 2 | 1 | 4 | 3 | 2 | 1 | Improvement suggestions |
| Overall evaluation of the program | | | | | | | | | |
| Duration | | | | | | | | | |
| Frequency | | | | | | | | | |
| Intensity | | | | | | | | | |
| Time | | | | | | | | | |
| Content of warm- up | | | | | | | | | |
| Content of physical training | | | | | | | | | |
| Content of cool down | | | | | | | | | |
| Sets and reps | | | | | | | | | |
| Rest time | | | | | | | | | |

#### **4 Outcome Measures**

## 4.1 Lower limb explosive power:

Countermovement jumps: experimenters test using either arm swing or crossed hips (without any arm swing) while performing vertical longitudinal jumps on a smart jumping mat. The experimenter in this research uses a cross-legged waist when performing both the pre-test and post-test. The Smart Jump Pad in this research has been performed to measure the performance of the CMJ by providing signals from the platform in an iPad 7,5 IOS 12.1.1). When the test equipment is ready, under the direction of the test administrator, the experimenter stands on the Smart Jump Mat and performs a vertical longitudinal jump. The experimenter jumps to the best of their ability and each jump was automatically recorded on the iPad. Each participant jumped three times, and the best jump results are selected for data analysis in this research.(Meszler et al., 2019)

۰



**Stangding long jumps:** Measure the distance of the standing long jump with a measuring tape.

Participants stand slightly apart in front of the jump line, bend their knees, and move their arms backwards, then swing their arms and jump as far as possible; Stand on both feet while maintaining an upright position; Conduct two tests. Record the best score from two tests with an accuracy of 1 centimeter (Ambroży et al., 2022).



**20m-sprint :** Use a stopwatch to record the duration of the participants' 30 m sprint.

Set cones at 0 and 20 meters along a straight line. Participants place their toes on the starting line or behind the starting line, start from a stationary position, and sprint at maximum speed over the cone at a distance of 20 meters before safely slowing down (Fischetti et al., 2018).



### 4.2 Latin Dance Performance

Using a video camera, a recorded video of the Cha Cha Gold Medal solo routine is send to the 6 judges, and the pre- and post-tests need to be rated using the same criteria 'the Latin Dance Technical Quality Elements of WDSF2.1 Evaluation System' Objectively assess posture, balance, footwork, preparation-movement-reduction, spinning and rotation, dynamic performance, and line extension (pei, 2023).

**Table 5 Scoring Standards for the Qualities of Cha-cha-cha Dancing Skills** 

| Indictors | Very excellent. (10 points) | excellent (8 points) | Above average (6 points) |
|---|---|---|---|
| Posture | Requires the ability to adopt and maintain correct posture during dynamic movement and, with minimal effort, to consciously demonstrate spatial transition postures. | It can drive the entire body to be integrated into the pose, so that the gesture blends with the posture. | The body, in static or dynamic motion, has a well-balanced body structure that includes the head, shoulders, chest, hips, legs, and feet. |
| Balance | Static: the line of gravity can be reconstructed after dynamic balance movement; Dynamic: can be used naturally and smoothly to generate three-dimensional movement effects, to realize the balance and effect of dance. | Static: can keep its own gravity in the extension line; Dynamic: the use of correct force to achieve dance balance, producing three-dimensional effects | Static: maintains the line of gravity from head to toe; Dynamic: maintaining balance while moving. |
| Footwork | Control of the spine through the flow of the steps and the transition between centers of gravity to complete the footwork. | Ability to properly utilize foot technique, connecting the necessary foot pressures and hip and body movements. | Ability to properly utilize foot technique. |
| Preparation-movement-reduction | The ability to perform the full range of motion with a natural and smooth transition from one movement to the next. | It is possible to make the transition<br>from one movement to another<br>during the performance of a<br>complete movement. | Most of the articulated pre-reduction from movement to movement can be accomplished when performing full movements. |
| Spinning and rotation | Maximize the use of centripetal and centrifugal forces in rotating and turning motions. | It is possible to combine the sagittal plane with the coronal plane when accomplishing rotational and turning. movements. | Ability to combine the sagittal and coronal planes most of the time when completing rotational and turning maneuvers |
| Dynamic performance | Precise use and maximization of power generation in dance movements. | Precise use of power in dance movements | Precise application of power in most dance movements |
| Line extension | Maintains the lines and extensions of all body parts in both static and dynamic situations. | Maintains most body lines and extensions in both static and dynamic situations. | Maintains a portion of the body line and extends the line in both static and dynamic situations. |

## **Table 6 Outcome Measurement Information**

| Test Name | Outcome<br>Measure | Measure Method | Instrument | Unit | Suggestions |
|---|---|---|---|---|---|
| | Countermo<br>vement<br>jumps | Recorded maximum altitude | Smart jump<br>mats, iPad | Centimeters (cm) | |
| Explosive power | Stangding long jumps | Measure the distance of the standing long jump with a measuring tape. | Measuring tape | Centimeters (cm) | |
| | 20m-sprint | Use a stopwatch to record the duration of the participants' 20 m sprint. | Stopwatch | Seconds | |
| Posture | 6 Experts | Recording<br>cha-cha-cha solo gold<br>medal moves, expert<br>scoring | M120<br>high-speed<br>camera | scores | |
| Balance | 6 Experts | Recording<br>cha-cha-cha solo gold<br>medal moves, expert<br>scoring | M120<br>high-speed<br>camera | scores | |
| Footwork | 6 Experts | Recording<br>cha-cha-cha solo gold<br>medal moves, expert<br>scoring | M120<br>high-speed<br>camera | scores | |
| Preparation-movement -reduction | 6 Experts | Recording<br>cha-cha-cha solo gold<br>medal moves, expert<br>scoring | M120<br>high-speed<br>camera | scores | |
| Spinning and rotation | 6 Experts | Recording<br>cha-cha-cha solo gold<br>medal moves, expert<br>scoring | M120<br>high-speed<br>camera | scores | |
| Dynamic performance | 6 Experts | Recording<br>cha-cha-cha solo gold<br>medal moves, expert<br>scoring | M120<br>high-speed<br>camera | scores | |
| Line extension | 6 Experts | Recording cha-cha-cha solo gold medal moves, expert scoring | M120<br>high-speed<br>camera | scores | |

## **5 Questionnaire information**

This questionnaire adopts a 5-point Likert scale, with 1-5 representing increasing support (1=strongly disagree; 2=disagree; 3=not necessarily; 4=agree; 5=strongly agree). Please score the intervention program. If there is other content, you can add them and indicate the name. After reading the questionnaire, please rate the following aspects and tick " $\sqrt{}$ " on the corresponding rating scale.

**Table 7 Expert Evaluation Form for Outcome Measurement** 

| Туре | Measurement Method | Rele | vance | ) | Clarity | | | | Improvement suggestions |
|---|---|---|---|---|---|---|---|---|---|
| | Measurement Method | 3 | 2 | 1 | 4 | 3 | 2 | 1 | |
| | Countermovement jumps | | | | | | | | |
| Explosive power | Stangding long jumps | | | | | | | | |
| | 20m-sprint | | | | | | | | |
| | Posture | | | | | | | | |
| | Balance | | | | | | | | |
| | Footwork | | | | | | | | |
| Latin dance performance | Preparation-movement-reduction | | | | | | | | |
| | Spinning and rotation | | | | | | | | |
| | Dynamic performance | | | | | | | | |
| | Line extension | | | | | | | | |

#### **6 References**

- Angioi, M., Metsios, G., Twitchett, E. A., Koutedakis, Y., & Wyon, M. (2012). Effects of supplemental training on fitness and aesthetic competence parameters in contemporary dance: a randomised controlled trial. Med Probl Perform Art, 27(1), 3-8.
- De La Cruz-Torres, B., Barrera-García-Martín, I., & Albornoz-Cabello, M. (2019). Immediate effects of ultrasound-guided percutaneous neuromodulation versus physical exercise on performance of the flexor hallucis longus muscle in professional dancers: A randomised clinical trial. Acupuncture in Medicine, 37(2), 91-97.
- Dowse, R. A., McGuigan, M. R., & Harrison, C. (2020). Effects of a resistance training intervention on strength, power, and performance in adolescent dancers. The Journal of Strength & Conditioning Research, 34(12), 3446-3453.
- Hutt, K., & Redding, E. (2014). The effect of an eyes-closed dance-specific training program on dynamic balance in elite pre-professional ballet dancers: a randomized controlled pilot study. Journal of Dance Medicine & Science, 18(1), 3-11.
- Karim, A., Roddey, T., Mitchell, K., Ortiz, A., & Olson, S. (2019). Immediate Effect of Whole Body Vibration on Sauté Height and Balance in Female Professional Contemporary Dancers: A Randomized Controlled Trial. Journal of Dance Medicine & Science, 23(1), 3-10.
- Kim, G., Kim, H., Kim, W. K., & Kim, J. (2017). Effect of stretching-based rehabilitation on pain, flexibility and muscle strength in dancers with hamstring injury: a single-blind, prospective, randomized clinical trial. The journal of sports medicine and physical fitness, 58(9), 1287-1295.
- Ko, M. G., Lee, M. M., & Song, C. H. (2020). A comparison of the effects of different stretching methods on flexibility, muscle activity, and pain threshold in ballet dancers; a preliminary randomized controlled trial. Journal of Bodywork and Movement Therapies, 24(4), 354-360.
- Kolokythas, N., Metsios, G. S., Galloway, S. M., Allen, N., & Wyon, M. A. (2022). Neuromuscular Training in Pre-Professional Ballet Dancers: A Feasibility Randomized Controlled Trial. Journal of Dance Medicine & Science, 26(3), 181-190.
- Koutedakis, Y., Hukam, H., Metsios, G., Nevill, A., Giakas, G., Jamurtas, A., & Myszkewycz, L. (2007). The effects of three months of aerobic and strength training on selected performance-and fitness-related parameters in modern dance students. The Journal of Strength & Conditioning Research, 21(3), 808-812.
- Koutedakis, Y., & Sharp, N. C. (2004). Thigh-muscles strength training, dance exercise, dynamometry, and anthropometry in professional ballerinas. The Journal of Strength & Conditioning Research, 18(4), 714-718.
- Liu, Y., & Wang, Y. (2024). Study on the effect of blood flow restriction training combined with IASTAM on ankle strength and function intervention in athletes with chronic ankle instability in sport dance events. BMC Sports Science, Medicine and Rehabilitation, 16(1), 1-17.
- Marshall, L. C., & Wyon, M. A. (2012). The effect of whole-body vibration on jump height and active range of movement in female dancers. The Journal of Strength & Conditioning Research, 26(3), 789-793.

- Moro, T., Marcolin, G., Bianco, A., Bolzetta, F., Berton, L., Sergi, G., & Paoli, A. (2020). Effects of 6 Weeks of Traditional Resistance Training or High Intensity Interval Resistance Training on Body Composition, Aerobic Power and Strength in Healthy Young Subjects: A Randomized Parallel Trial. Int J Environ Res Public Health, 17(11).
- Huang, H., Huang, W.-Y., & Wu, C.-E. (2023). The effect of plyometric training on the speed, agility, and explosive strength performance in elite athletes. Applied Sciences, 13(6), 3605.
- Ramírez-Campillo, R., Álvarez, C., Henríquez-Olguín, C., Baez, E. B., Martínez, C., Andrade, D. C., & Izquierdo, M. (2014). Effects of plyometric training on endurance and explosive strength performance in competitive middle-and long-distance runners. The Journal of Strength & Conditioning Research, 28(1), 97-104.
- Ramírez-Campillo, R., Andrade, D. C., & Izquierdo, M. (2013). Effects of plyometric training volume and training surface on explosive strength. The Journal of Strength & Conditioning Research, 27(10), 2714-2722.
- Du, M. (2020). Effects of plyometric training on lower extremity explosive strength and athletic performance in adolescent Latin dancers (Master Dissertation). Beijing Sport University, Bei Jing.
- Chen, L., Zhang, Z., Huang, Z., Yang, Q., Gao, C., Ji, H., ... & Li, D. (2023). Meta-analysis of the effects of plyometric training on lower limb explosive strength in adolescent athletes. International journal of environmental research and public health, 20(3), 1849.
- Pei J, J. (2023). Effects of plyometric training on the technical quality of movement in 15-16 year old female cha-cha dancers (Master Dissertation), Shanghai University of Sport, Shang Hai.